CLINICAL TRIAL: NCT04903587
Title: The Prevalence Of Gonadal Changes In Patients With Congenital Adrenal Hyperplasia
Brief Title: Gonadal Changes In Congenital Adrenal Hyperplasia Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: US and MRI in CAH patients
Record Dates: First submitted 2021-05-23; First posted 2021-05-26 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-05

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasonography and MRI — Abdominal Ultrasonography and axial MRI

SUMMARY:
To detect the prevalence of gonadal changes by US among the patients with CAH.

* assess the patients' radiological findings in relation to their hormonal profile.
* early management and prevention of complications resulting from possible gonadal dysfunction.

DETAILED DESCRIPTION:
Several factors contribute to the impaired fertility in CAH patients, such as androgen excess, adrenal progesterone hypersecretion and adrenal rest tumours (ARTs). ARTs are derived from ectopic adrenal cells that migrated to the gonads in foetal life, and their growth is under control of adrenocorticotropic hormone (ACTH) and angiotensin II .

The common cause of infertility in males with CAH is testicular adrenal rest tumours (TARTs) , which have been well documented in CAH male patients, with an incidence up to 94%. They could be easily imaged by US and MRI studies. TARTs are associated with the risk of seminal duct obstruction, leading to azoospermia and permanent damage of the surrounding testicular tissue. TARTs can present as single nodules , and as multiple nodules in 16% of patients. Increasing the dosage of hormone therapy can cause early TARTs lesions to shrink or completely resolve, while advanced lesions may require surgical removal .

High prevalence of impaired fertility is not restricted to men; as it was reported also in women with CAH. Androgen excess is usually implicated in girls and women with CAH for whom medical treatment is unavailable or who are noncompliant with their therapy . Adrenal androgens act either directly or through the dysfunction caused at the hypothalamic pituitary axis. Interestingly, ovarian hyperandrogenism could occur even when CAH is well controlled on glucocorticoid therapy .

Females with CAH may become infertile for several reasons, such as chronic anovulation, which was demonstrated in up to 50% of the patients with non-classic CAH . Bilateral enlarged ovaries, bilateral ovarian cysts, and ovarian adrenal rest tumour (OART) may also occur and can be detected by US. OART impairs ovarian function in CAH females by displacing normal ovarian tissue and by locally producing steroids, which interfere with normal ovarian function. It should be considered when ovarian masses are detected. If detected early enough and glucocorticoid therapy is received, it is possible that it will decrease in size following suppression of ACTH levels. Polycystic ovary syndrome (PCOS) is another common condition associated with hyperandrogenism. The prevalence of PCOS is increased in women with both classical and non-classical CAH. The association of CAH with ultrasonically detected PCOS was confirmed in 83%, 40% and 3% of the adult patients, postpubertal girls and pre and peripubertal girls respectively .

Under treatment of ARTs, PCOS and other gonadal comorbidities negatively influences the quality of life as well as sexual outcomes in patients with CAH. Besides, recognizing these conditions and identifying characteristic US features of gonadal dysfunction is important, so as to avoid misdiagnosing them as malignancies, which can lead to unnecessary interventions.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with CAH between five and 16 years of age will be asked to participate in this cross sectional study.
* Compliant patients with regular follow up.

Exclusion Criteria:

* Presence of other endocrinal diseases or chronic conditions.
* Female patients with ovulatory dysfunction from other causes including thyroid dysfunction and hyperprolactinemia.
* Male patients with other diseases causing impairment of gonadal capacity.

Ages: 5 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: all patients diagnosed with congenital adrenal hyperplasia (CAH)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
prevalence of gonadal changes in CAH patients | baseline
  By using US and MRI to detect the finding in gonades in CAH patients

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] Dumic M, Duspara V, Grubic Z, Oguic SK, Skrabic V, Kusec V. Testicular adrenal rest tumors in congenital adrenal hyperplasia-cross-sectional study of 51 Croatian male patients. Eur J Pediatr. 2017 Oct;176(10):1393-1404. doi: 10.1007/s00431-017-3008-7. Epub 2017 Sep 6. PMID 28879515
- [Background] Chen HD, Huang LE, Zhong ZH, Su Z, Jiang H, Zeng J, Liu JC. Ovarian Adrenal Rest Tumors Undetected by Imaging Studies and Identified at Surgery in Three Females with Congenital Adrenal Hyperplasia Unresponsive to Increased Hormone Therapy Dosage. Endocr Pathol. 2017 Jun;28(2):146-151. doi: 10.1007/s12022-016-9461-4. PMID 28032206